CLINICAL TRIAL: NCT01537666
Title: Phase I, Reference-controlled, Dose Escalating Study to Examine the Pharmacokinetics and Safety of AeroVanc Inhalation Powder.
Brief Title: Inhaled Vancomycin Tolerability, Safety and Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Collaborators: INC Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAV005-01
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Aerovanc 16 mg in healthy volunteers (Experimental)
  Interventions: Drug: AeroVanc
- AeroVanc 32 mg in healthy volunteers (Experimental)
  Interventions: Drug: AeroVanc
- AeroVanc 80 mg in healthy volunteers (Experimental)
  Interventions: Drug: AeroVanc
- IV vancomycin in healthy volunteers (Active Comparator)
  Interventions: Drug: IV vancomycin hydrochloride
- AeroVanc 32 mg in CF patients (Experimental)
  Interventions: Drug: AeroVanc
- AeroVanc 80 mg in CF patients (Experimental)
  Interventions: Drug: AeroVanc

INTERVENTIONS:
Drug: AeroVanc — Vancomycin hydrochloride dry powder for inhalation
  Arms: AeroVanc 32 mg in CF patients; AeroVanc 32 mg in healthy volunteers; AeroVanc 80 mg in CF patients; AeroVanc 80 mg in healthy volunteers; Aerovanc 16 mg in healthy volunteers
Drug: IV vancomycin hydrochloride — Vancomycin hydrochloride solution for intravenous administration
  Arms: IV vancomycin in healthy volunteers

SUMMARY:
The study is carried out to evaluate the safety, tolerability and pharmacokinetics of AeroVanc inhalation powder in healthy volunteers, and in patients with cystic fibrosis.

DETAILED DESCRIPTION:
The study has three main objectives:

* To evaluate the safety, and tolerability of AeroVanc inhalation powder in healthy volunteers, and in patients with CF.
* To determine the systemic bioavailability of vancomycin in healthy volunteers following single dose pulmonary administration of 16 mg, 32 mg, and 80 mg doses of AeroVanc in comparison with a 250 mg dose of vancomycin administered intravenously.
* To estimate the lung sputum concentrations of vancomycin in patients with cystic fibrosis (CF) following single dose pulmonary administration of 32 mg and 80 mg doses of AeroVanc.

ELIGIBILITY:
Inclusion Criteria Healthy Volunteers:

1. Healthy male volunteers between 18 and 50 years of age inclusive.
2. Able to communicate with site personnel and to understand and voluntarily sign the Informed Consent Form.
3. Able and willing to comply with the Protocol, including availability for all scheduled study visits.
4. Body Mass Index (BMI) of 20 to 30 kg/m2 inclusive, and weight between 60-90 kg inclusive.
5. No clinically significant abnormalities at screening determined by medical history, physical examination, blood chemistry, hematology, urinalysis, and 12-lead ECG. Negative urine screen for drugs of abuse and negative alcohol breath test at Screening and prior to dosing.
6. Negative human immunodeficiency virus (HIV) and Hepatitis B and Hepatitis C screening test results.
7. Spirometry (forced expiratory volume in 1 second (FEV1)) value at screening greater than 75% of predicted age-adjusted value.

Exclusion Criteria Healthy Volunteers:

1. A history of pulmonary or other disorder likely to influence drug absorption.
2. Evidence or suspicion of clinically significant respiratory, renal, hepatic, central nervous system, cardiovascular or metabolic dysfunction.
3. A history of previous allergies or sensitivity to vancomycin, or other component(s) of the study drug or reference drug.
4. Smokers (ex-smokers who quit smoking must have a one year period of not smoking prior to the study drug administration).
5. Respiratory tract infection within the last two weeks prior to the first study drug administration.
6. Treatment with any prescription medication and/or over-the-counter (OTC) products including vitamins or mineral supplements within 48 hours before Investigational Product administration.
7. Vaccination within one month before the study drug administration.
8. Systolic blood pressure <110 mmHg or >150 mmHg inclusive or diastolic blood pressure <60 mmHg or >90 mmHg inclusive.
9. A history of drug or alcohol abuse.
10. Participation in a clinical study within three months on Investigational Product administration.
11. Donation of blood or plasma within three months of Investigational Product administration.
12. Any other condition which in the view of the Investigator is likely to interfere with the study or put the subject at risk.

Inclusion Criteria CF Patients:

1. Able to communicate with site personnel and to understand and voluntarily sign the Informed Consent Form.
2. Able and willing to comply with the protocol, including availability for all scheduled study visits.
3. Have a confirmed diagnosis of cystic fibrosis (by two established methods, e.g. positive sweat chloride value ≥ 60 mEq/L, nasal potential difference test, and/or genotype with two identifiable mutations consistent with CF, accompanied by one or more clinical features consistent with the CF phenotype).
4. Be aged ≥ 18 years old
5. Have FEV1 >40 % of predicted
6. Be able to perform all the techniques necessary to measure lung function
7. No liver enzymes increased by more than twice the upper limit of normal
8. Ability to spontaneously produce bronchial sputum daily

Inclusion Criteria CF Patients:

1. Administration of any investigational drug or device within 28 days of Screening and within six half-lives of the investigational drug.
2. Oral corticosteroids in doses exceeding 10 mg per day or 16 mg every other day.
3. History of sputum culture or throat swab culture yielding B. cepacia in the previous two years.
4. History of positive MRSA culture, or sputum culture positive for MRSA at screening.
5. Current daily continuous oxygen supplementation or requirement for more than 2 L/min at night.
6. A history of previous allergies or sensitivity to vancomycin, or other component(s) of the study drug.
7. Changes in antimicrobial, bronchodilator, anti-inflammatory or corticosteroid medications within 7 days prior to Screening.
8. Changes in physiotherapy technique or schedule within 7 days prior to Screening.
9. History of lung transplantation.
10. A chest X-Ray at Screening or within the previous 90 days of Screening, with abnormalities indicating a significant acute finding (e.g., lobar infiltrate and atelectasis, pneumothorax, or pleural effusion).
11. Positive pregnancy test. All women of childbearing potential will be tested.
12. Female of childbearing potential who is lactating or is not practicing acceptable method of birth control (e.g., hormonal or barrier methods, or intrauterine device).
13. Findings at Screening that, in the investigator's opinion, would compromise the safety of the subject or the quality of the study data.
14. History of severe cough/bronchospasm upon inhalation of dry powder inhalation product.
15. Considered "terminally ill" or eligible for lung transplantation.
16. Have had a significant episode of hemoptysis (>60 mL) in the three months prior to enrolment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Mater Adult Hospital, Brisbane, Queensland
  - Linear Clinical Research Ltd., Perth, Western Australia

RESULTS

PARTICIPANT FLOW:
Groups:
- Aerovanc 16 mg (Subset IV Vancomycin) in Healthy Volunteers; AeroVanc 32 mg (Subset IV Vancomycin) in Healthy Volunteers; AeroVanc 80 mg (Subset IV Vancomycin) in Healthy Volunteers: AeroVanc : Vancomycin hydrochloride dry powder for inhalation (N=6)/ Subset received IV vancomycin hydrochloride : Vancomycin hydrochloride solution for intravenous administration (N=2 from this group, 6 overall)
- AeroVanc 32 and 80 mg in CF Patients: AeroVanc : Vancomycin hydrochloride dry powder for inhalation
Period: Overall Study
Arm/Group | Aerovanc 16 mg (Subset IV Vancomycin) in Healthy Volunteers | AeroVanc 32 mg (Subset IV Vancomycin) in Healthy Volunteers | AeroVanc 80 mg (Subset IV Vancomycin) in Healthy Volunteers | AeroVanc 32 and 80 mg in CF Patients
Started | 6 (2 of these 6 also received a single 250 mg IV dose of vancomycin at least 72 hours after AeroVanc.) | 6 (2 of these 6 also received a single 250 mg IV dose of vancomycin at least 72 hours after AeroVanc.) | 6 (2 of these 6 also received a single 250 mg IV dose of vancomycin at least 72 hours after AeroVanc.) | 7 (5 of 7 patients received a 32 mg dose of AeroVanc followed by a dose of 80 mg at least 1 week later.)
Completed | 6 | 6 | 6 | 7 (1 patient withdrew after a 32 mg dose and was replaced by a patient who only received an 80 mg dose.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerovanc 16 mg (Subset IV Vancomycin) in Healthy Volunteers | AeroVanc 32 mg (Subset IV Vancomycin) in Healthy Volunteers | AeroVanc 80 mg (Subset IV Vancomycin) in Healthy Volunteers | AeroVanc 32 and 80 mg in CF Patients | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 7 | 25
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (10.5) | 24.7 (3.7) | 22.2 (2.8) | 29.7 (7.8) | 26.3 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 3 | 3
  Male | 6 | 6 | 6 | 4 | 22
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 6 | 6 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability - Number of Participants With Treatment Emergent Adverse Events (TEAEs = Adverse Events That Started During or After the First Dose of Study Drug)
Description: Each participant was monitored regularly for Adverse Events (AEs) throughout the study. The Investigator or designee enquired about AEs by asking participants non-leading questions such as: "How do you feel?" or "Have you had any (other) medical problems since your last visit/assessment?" Additionally, several safety procedures (physical examinations, vital signs, safety laboratory tests, 12-lead ECGs, and spirometry) were conducted on participants at regular intervals. All AEs reported spontaneously by participants or in response to questioning or observation by the Investigator, including those related to safety procedures, were recorded. For each AE, the Investigator recorded the following assessments: seriousness, severity (Mild, Moderate, or Severe), and relationship to study drug (Not Related, Remote, Possible, Probable, or Highly Probable). AEs were considered drug-related if given a relationship of Possible, Probable, or Highly Probable.
Time Frame: Healthy volunteers = 2 weeks; CF Patients = 1 week
Population: All 18 healthy volunteers who received single doses of AeroVanc, 6 of which also received a single dose of IV vancomycin. All 7 Cystic Fibrosis patients who received at least one single dose of AeroVanc.
Measure: Number; unit: participants
Groups:
- AeroVanc 16 mg in Healthy Volunteers: Single inhaled dose of 16 mg AeroVanc in health volunteers.
- AeroVanc 32 mg in Healthy Volunteers: Single inhaled dose of 32 mg AeroVanc in health volunteers.
- AeroVanc 80 mg in Healthy Volunteers: Single inhaled dose of 80 mg AeroVanc in health volunteers.
- IV Vancomycin 250 mg in Healthy Volunteers: Single IV dose of Vancomycin 250 mg in Healthy Volunteers. Group comprised of 2 subjects from each of the AeroVanc in Healthy Volunteers groups.
- AeroVanc 32 mg in Cystic Fibrosis Patients: Single inhaled dose of 32 mg AeroVanc. One patient withdrew after receiving a 32 mg dose and was replaced with a patient who only received an 80 mg dose.
- AeroVanc 80 mg in Cystic Fibrosis Patients: Single inhaled dose of 80 mg AeroVanc. One patient withdrew after receiving a 32 mg dose and was replaced with a patient who only received an 80 mg dose.
Arm/Group | AeroVanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | IV Vancomycin 250 mg in Healthy Volunteers | AeroVanc 32 mg in Cystic Fibrosis Patients | AeroVanc 80 mg in Cystic Fibrosis Patients
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6
participants
  Total with at least one TEAE | 2 | 5 | 2 | 2 | 6 | 5
  Subset of total with drug-related TEAEs | 2 | 3 | 2 | 1 | 4 | 4
  Subset of total with severe TEAEs | 0 | 0 | 0 | 0 | 1 | 0
  Subset of total with severe, drug-related TEAEs | 0 | 0 | 0 | 0 | 0 | 0
  Subset of total with serious TEAEs | 0 | 0 | 0 | 0 | 1 | 0
  Subset of total with serious, drug-related TEAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Plasma Pharmacokinetics - Elimination Half Life (t½)
Description: Blood samples were obtained from the healthy volunteers to evaluate systemic pharmacokinetics of vancomycin after a single dose administration of AeroVanc or a single dose of IV vancomycin.
  Half-life is the time it takes for the concentration of drug to decline by 50%.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: All healthy volunteers (N=18) who received a single 16, 32, or 80 mg inhaled dose of AeroVanc. Subset (N=6 comprised of 2 patients from each of the AeroVanc groups) who received a single 250 mg IV dose of vancomycin.
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Aerovanc 16 mg in Healthy Volunteers; AeroVanc 32 mg in Healthy Volunteers; AeroVanc 80 mg in Healthy Volunteers: AeroVanc : Vancomycin hydrochloride dry powder for inhalation
- IV Vancomycin 250 mg in Healthy Volunteers: IV vancomycin hydrochloride : Vancomycin hydrochloride solution for intravenous administration
Arm/Group | Aerovanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | IV Vancomycin 250 mg in Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 8.454 (2.017) | 8.648 (0.530) | 8.044 (1.296) | 7.226 (1.128)

3. Secondary Outcome: Plasma Pharmacokinetics - Time to Reach the Maximum Plasma Concentration (Tmax)
Description: Blood samples were obtained from the healthy volunteers to evaluate systemic pharmacokinetics of vancomycin after a single dose administration of AeroVanc or a single dose of IV vancomycin.
  Tmax is the time it takes to reach the maximum plasma concentration of a drug.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Aerovanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | IV Vancomycin 250 mg in Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hours | 2.083 (0.801) | 1.833 (0.606) | 1.333 (0.408) | 0.917 (0.204)

4. Secondary Outcome: Plasma Pharmacokinetics - Maximum Plasma Concentration (Cmax)
Description: Blood samples were obtained from the healthy volunteers to evaluate systemic pharmacokinetics of vancomycin after a single dose administration of AeroVanc or a single dose of IV vancomycin.
  Cmax is the maximum observed concentration of a drug.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Aerovanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | IV Vancomycin 250 mg in Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng/ml | 108.82 (33.16) | 231.50 (89.64) | 617.83 (230.03) | 10028.33 (1767.69)

5. Secondary Outcome: Plasma Pharmacokinetics - Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUCt)
Description: Blood samples were obtained from the healthy volunteers to evaluate systemic pharmacokinetics of vancomycin after a single dose administration of AeroVanc or a single dose of IV vancomycin.
  AUCt is a way of expressing the total amount of drug exposure over a specified time period.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Aerovanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | IV Vancomycin 250 mg in Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/ml | 1209.644 (237.696) | 2379.790 (975.410) | 6257.858 (1506.939) | 41027.792 (2696.013)

6. Secondary Outcome: Plasma Pharmacokinetics - Area Under the Plasma Concentration-time Curve From Time 0 to Infinite Time (AUCinf)
Description: Blood samples were obtained from the healthy volunteers to evaluate systemic pharmacokinetics of vancomycin after a single dose administration of AeroVanc or a single dose of IV vancomycin.
  AUCinf is a way of estimating the total amount of drug exposure over an infinite time period.
Time Frame: Pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Aerovanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | IV Vancomycin 250 mg in Healthy Volunteers
Number analyzed (Participants) | 6 | 6 | 6 | 6
h*ng/ml | 1461.407 (257.189) | 3051.12 (959.14) | 7135.735 (1457.921) | 44356.356 (3623.420)

7. Secondary Outcome: Lung Pharmacokinetics - Maximum Sputum Concentration (Cmax)
Description: Sputum samples were obtained from the patients with cystic fibrosis to evaluate lung pharmacokinetics of vancomycin after a single dose administration of AeroVanc.
  Cmax is the maximum observed concentration of a drug.
Time Frame: 1, 8 and 24 hours post-dose
Population: All CF patients who received a 32 mg dose of AeroVanc followed at least one week later by an 80 mg dose of AeroVanc (N=5). One patient withdrew after receiving a 32 mg dose and was replaced with a patient who only received an 80 mg dose.
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | AeroVanc 32 mg in Cystic Fibrosis Patients | AeroVanc 80 mg in Cystic Fibrosis Patients
Number analyzed (Participants) | 6 | 6
µg/ml | 95.775 (171.544) | 269.17 (510.98)

8. Secondary Outcome: Lung Pharmacokinetics - Minimum Sputum Concentration (Cmin)
Description: Sputum samples were obtained from the patients with cystic fibrosis to evaluate lung pharmacokinetics of vancomycin after a single dose administration of AeroVanc.
  Cmin is the minimum observed concentration of a drug.
Time Frame: 1, 8 and 24 hours post-dose
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: µg/ml
Arm/Group | AeroVanc 32 mg in Cystic Fibrosis Patients | AeroVanc 80 mg in Cystic Fibrosis Patients
Number analyzed (Participants) | 6 | 6
µg/ml | 3.050 (3.679) | 7.990 (8.066)

ADVERSE EVENTS:
Time Frame: All 25 subjects enrolled received at least part of their allocated study treatments and are included in the safety population. All subjects received their allocated dose, and in Part 2 of the study, 5 subjects received both the 32 mg and 80 mg doses.
Description: AEs were grouped by system organ class and summarized by dose level at the time of onset of the AE. All AE summaries are restricted to TEAEs, defined as AEs that began on or after the start of study drug. AEs without an onset date or time were excluded from the summary tables as it was not possible to allocate to a particular treatment.
Groups:
- IV Vancomycin 250 mg in Healthy Volunteers: Comprised of 2 patients from each of the AeroVanc in Healthy Volunteer groups.
Arm/Group | AeroVanc 16 mg in Healthy Volunteers | AeroVanc 32 mg in Healthy Volunteers | AeroVanc 80 mg in Healthy Volunteers | AeroVanc 32 mg in Cystic Fibrosis Patients | AeroVanc 80 mg in Cystic Fibrosis Patients | IV Vancomycin 250 mg in Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 5/6 | 2/6 | 6/6 | 5/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroVanc 16 mg in Healthy Volunteers (N=6) | AeroVanc 32 mg in Healthy Volunteers (N=6) | AeroVanc 80 mg in Healthy Volunteers (N=6) | AeroVanc 32 mg in Cystic Fibrosis Patients (N=6) | AeroVanc 80 mg in Cystic Fibrosis Patients (N=6) | IV Vancomycin 250 mg in Healthy Volunteers (N=6)
AGGRAVATED RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroVanc 16 mg in Healthy Volunteers (N=6) | AeroVanc 32 mg in Healthy Volunteers (N=6) | AeroVanc 80 mg in Healthy Volunteers (N=6) | AeroVanc 32 mg in Cystic Fibrosis Patients (N=6) | AeroVanc 80 mg in Cystic Fibrosis Patients (N=6) | IV Vancomycin 250 mg in Healthy Volunteers (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot at any time during or after the Study make any announcement, oral presentation or publication relating to the Study, or any of the methods, results of, or conclusions from, the Study without the prior written consent of the Sponsor.